CLINICAL TRIAL: NCT05400694
Title: The Sensory and Metabolic Effects of Functional and Value-Added Dairy Products
Brief Title: Functional and Value-Added Dairy Products and Blood Glucose Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Saint Vincent University (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Bohdan Luhovyy, Associate Professor, Mount Saint Vincent University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-202-02
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Blood Glucose, High; Metabolic Disease; Overweight and Obesity
Keywords: Sugar intake; Sweeteners; Milk Proteins; Diabetes; Obesity; Sweetened food products; Chocolate milk; Blood glucose; Insulin; Satiety; Food Intake; Casein; Whey protein
MeSH Terms: conditions — Metabolic Diseases; Overweight; Obesity; Diabetes Mellitus; Insulin Resistance | interventions — Food

STUDY DESIGN:
Who Masked: Participant
Masking Description: Treatments are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Chocolate milk (Experimental): Chocolate milk with reduced added sugar
  Interventions: Other: Food
- Chocolate milk with whey protein (Experimental): Chocolate milk with reduced added sugar and added whey protein
  Interventions: Other: Food
- Chocolate milk with casein (Experimental): Chocolate milk with reduced added sugar and added casein
  Interventions: Other: Food
- Chocolate milk with alpha-lactalbumin (Experimental): Chocolate milk with reduced added sugar and added alpha-lactalbumin
  Interventions: Other: Food
- Chocolate milk with glycomacropeptide (Experimental): Chocolate milk with reduced added sugar and added glycomacropeptide
  Interventions: Other: Food

INTERVENTIONS:
Other: Food — Dairy products with reduced sugar content

SUMMARY:
Milk proteins possess multiple biological activities including their effect on blood glucose control, satiety and energy intake. The design of functional food products with added milk protein fractions has many challenges related to their inferior sensory properties. Chocolate milk presents the universal vehicle for added milk protein fractions that might partially mask their sensory characteristics. However, commercially produced chocolate milk has a significant amount of added sugar. This project will investigate the properties of a value-added dairy product (chocolate milk with reduced sugar content) enriched with individual milk protein fractions on characteristics of blood glucose control, satiety and energy intake in young healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* 19-35 y males and females, non-smokers

Exclusion Criteria:

* having any diseases, irregular menses in females, smoking (all types), taking medications known to influence blood glucose control, skipping breakfast, and having emotional, or learning problems that would affect their ability to participate in the study as required. Individuals with known food allergies and lactose intolerance will be also excluded.

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Blood glucose | 0-120 minutes
  The concentration of blood glucose
Insulin | 0-120 minutes
  The concentration of insulin

SECONDARY OUTCOMES:
C-peptide | 0-120 minutes
  The concentration of C-peptide
Incretins, glucagon and amino acids | 0-120 minutes
  The concentration of incretins and glucagon
Satiety | 0-120 minutes
  The components of average subjective appetite including desire to eat, hunger, fullness, and a prospective food consumption measured with 100mm visual analogue scales.
Food Intake | 0 min, 120 minutes
  Energy intake with an ad libitum meat at 120 minutes
Thirst | 0-120 minutes
  The subjective perception of thirst measured with 100mm visual analogue scales containing the question "How thirsty do you feel?" and two statements on each pole of 100mm line: "Not thirsty at all" (0mm) and "As thirsty as I have ever felt" (100mm).
Physical comfort | 0-120 minutes
  The subjective feeling of wellness and gastrointestinal discomfort parameters including the feeling of nausea, stomach cramps, flatulency, diarrhea and a subjective feeling of wellness, each measured with 100mm visual analogue scales.
Food pleasantness | at 0 and 120 minutes
  The perception of pleasantness of the treatments (0 minutes) and a test meal (at 120 minutes) will be measured with 100mm visual analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: Bohdan Luhovyy, PhD, Principal Investigator — Mount Saint Vincent University
Locations (1):
- Mount Saint Vincent University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No